CLINICAL TRIAL: NCT05883852
Title: A Randomized Controlled, Phase III Trial in HER2-positive Lymph Node Positive Early Breast Cancer to Compare the Efficacy and Safety of Epriubin Plus Cyclophosphamide Followed by Docetaxel Plus Trastuzumab and Pertuzumab (EC-THP) Versus Docetaxel and Carboplatin Plus Trastuzumab and Pertuzumab (TCbHP) in the Adjuvant Treatment
Brief Title: EC-THP Versus TCbHP in HER2-positive Lymph Node Positive Early Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N055
Record Dates: First submitted 2023-05-20; First posted 2023-06-01 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: HER2 Positive Early Breast Cancer
MeSH Terms: interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A：TCbHP (Experimental): Docetaxel 75mg/m2 ivgtt d1+ carboplatin AUC=6 ivgtt d1+ trastuzumab first dose 8mg/kg (maintain 6mg/kg) d1 ivgtt d1+ Pertuzumab first dose 840mg (maintain 420mg) ivgtt d1, 3 weeks of treatment, a total of 6 courses. After the completion of chemotherapy, the dual-target therapy was continued for one year.
  Interventions: Drug: Docetaxel; Drug: carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- Arm B：EC-THP (Active Comparator): Epirubicin 90 mg/m2 ivgtt d1+ cyclophosphamide 600 mg/m2 iv d1, 3 weeks of treatment, a total of 4 courses; Docetaxel 100mg/m2 ivgtt d1+ trastuzumab first dose 8mg/kg (maintenance 6mg/kg) d1 ivgtt d1+ pertuzumab first dose 840mg (maintenance 420mg) ivgtt d1, 3 weeks of treatment, a total of 6 courses. After the completion of chemotherapy, the dual-target therapy was continued for one year.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Epirubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel — Docetaxel is a taxoid antineoplastic agent used in the treatment of breast cancer
Drug: carboplatin — Carboplatin is a DNA synthesis inhibitor which binds to DNA, inhibits replication and transcription and induces cell death.
  Arms: Arm A：TCbHP
Drug: Trastuzumab — Trastuzumab is a humanized monoclonal antibody derived from recombinant DNA,
Drug: Pertuzumab — Pertuzumab is a recombinant humanized monoclonal antibody that specifically binds to the extracellular dimerization domain (subdomain Ⅱ) of epidermal growth factor receptor 2(HER2).
Drug: Epirubicin — Epirubicin is an antineoplastic agent derived from doxorubicin.Epirubicin, like doxorubicin, exerts its antitumor effects by interference with the synthesis and function of DNA and is most active during the S phase of the cell cycle.
  Arms: Arm B：EC-THP
Drug: cyclophosphamide — An anticancer (antitumor or cytotoxic) chemotherapy drug that is classified as an alkylating agent. Alkylating agents are compounds that prevent the normal connection of the double helix chain by adding an alkyl group to the guanine base of the DNA molecule. It causes breaks in DNA strands, affecting the ability of cancer cells to proliferate.
  Arms: Arm B：EC-THP

SUMMARY:
compare the efficacy and safety of TCbHP and EC-THP regimen in HER2-positive breast cancer patients

DETAILED DESCRIPTION:
The objective of this study is to conduct a randomized controlled clinical study to compare the efficacy and safety of TCbHP and EC-THP regimen in HER2-positive breast cancer patients, so as to further optimize adjuvant chemotherapy regimen for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70；
* 0-1 for ECOG；
* Unilateral invasive carcinoma confirmed by histology (regardless of pathological type)；
* No gross or microscopic tumor remains after surgical resection；
* Early breast cancer, pathologically confirmed as HER2 positive; HER2 positive definition: Immunohistochemical HER2 3+ or FISH/CISH test positive (with amplification) is defined as HER2 positive；
* Postoperative pathological stage pT1-4N1-3M0；
* Did not receive neoadjuvant chemotherapy in the past；
* The longest period from surgery to randomization was not more than 8 weeks, and no adjuvant therapy had been received after surgery；
* No peripheral neuropathy；
* Good postoperative recovery, at least 1 week interval between operation；
* The major organs function normally, that is, meet the following criteria: (1) The standard of blood routine examination shall meet: HB ≥90 g/L (no blood transfusion within 14 days); ANC ≥1.5×109 /L; PLT ≥100×109 /L; (2) Biochemical examination should meet the following standards: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3 x ULN; Serum Cr ≤1.5×ULN；
* Contraception during treatment for women of reproductive age；
* Cardiac function: LVEF>50% for ultrasound examination；
* The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up。

Exclusion Criteria:

* Bilateral breast cancer or carcinoma in situ DCIS/LCIS；
* Have received chemotherapy for advanced disease；
* Transfer of any part；
* If any tumor >T4a (accompanied by skin invasion, mass adhesion fixation, inflammatory breast cancer)；
* Patients with clinical or imaging suspicion of malignancy on the opposite breast but not confirmed, requiring biopsy；
* Have received neoadjuvant therapy, including chemotherapy, radiotherapy and endocrine therapy；
* Malignant neoplasms (other than basal cell carcinoma of the skin and carcinoma in situ of the cervix), including contralateral breast cancer, within the previous 5 years；
* The patient has been enrolled in other clinical trials；
* Patients with severe systemic disease and/or uncontrolled infection were unable to be enrolled in the study；
* LVEF<50% (cardiac ultrasound)；
* Severe cardiovascular and cerebrovascular disease (e.g., unstable angina, chronic heart failure, uncontrolled hypertension >150/90mmgh, myocardial infarction or cerebrovascular accident) within 6 months prior to randomization；
* Known allergy to related drugs；
* Women of childbearing age refuse contraception during treatment and within 8 weeks after completion of treatment；
* Pregnant and lactating women；
* Those who tested positive for pregnancy before taking the drug after joining the trial；
* Mental illness, cognitive impairment, inability to understand the trial protocol and side effects, inability to complete the trial protocol and follow-up workers ；(systematic evaluation is required before trial enrollment)；
* Persons without personal freedom and independent capacity for civil conduct。

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 1406 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2031-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
iDFS | 5 years
  invasive Disease Free Survival

SECONDARY OUTCOMES:
DRFS | 5 years
  distant relapse free survival
OS | 5 years
  overall survival
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  Incidence of treatment-emergent adverse events adverse events according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China